CLINICAL TRIAL: NCT04290039
Title: A Randomized, Three-Sequence, Three-Period Crossover Study to Assess the Bioavailability and Pharmacokinetics of a Single Dose of Atropine Administered Sublingually in Healthy Adult Volunteers
Brief Title: Sublingual vs IV Atropine Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BP-C-19010
Record Dates: First submitted 2020-01-27; First posted 2020-02-28 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Toxic Effect of Organophosphate and Carbamate Insecticides
MeSH Terms: interventions — Atropine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low Dose Sublingual (Active Comparator): Atropine sulfate ophthalmic solution, USP 1% is a sterile topical anti-muscarinic indicated for cyclopegia, mydriasis, and penalization of the healthy eye in the treatment of amblyopia. Each mL of Atropine Sulfate Ophthalmic Solution USP, 1% contains active ingredient: atropine sulfate 10 mg equivalent to 8.3 mg of atropine. Inactive ingredients include benzalkonium chloride 0.1 mg (0.01%), dibasic sodium phosphate, edetate disodium, hypromellose (2910), monobasic sodium phosphate, hydrochloric acid and/or sodium hydroxide may be added to adjust pH (3.5 to 6.0), and water for injection, USP. Atropine Sulfate Ophthalmic Solution, USP 1% will be supplied in dropper bottles containing 2 mL.
  Each bottle will only be used to administer a single dose, to a single subject.
  Interventions: Drug: Atropine Sulfate Ophthalmic Solution
- High Dose Sublingual (Active Comparator): Atropine sulfate ophthalmic solution, USP 1% is a sterile topical anti-muscarinic indicated for cyclopegia, mydriasis, and penalization of the healthy eye in the treatment of amblyopia. Each mL of Atropine Sulfate Ophthalmic Solution USP, 1% contains active ingredient: atropine sulfate 10 mg equivalent to 8.3 mg of atropine. Inactive ingredients include benzalkonium chloride 0.1 mg (0.01%), dibasic sodium phosphate, edetate disodium, hypromellose (2910), monobasic sodium phosphate, hydrochloric acid and/or sodium hydroxide may be added to adjust pH (3.5 to 6.0), and water for injection, USP. Atropine Sulfate Ophthalmic Solution, USP 1% will be supplied in dropper bottles containing 2 mL.
  Each bottle will only be used to administer a single dose, to a single subject.
  Interventions: Drug: Atropine Sulfate Ophthalmic Solution
- Intravenous (IV) (Active Comparator): Atropine sulfate injection is indicated for temporary blockade of severe or life-threatening muscarinic effects, e.g., as an antisialagogue, an antivagal agent, an antidote for organophosphorus, carbamate, or muscarinic mushroom poisoning, and to treat symptomatic bradycardia.
  Atropine sulfate injection, USP,8mg/20mL (0.4 mg per mL) is a sterile, nonpyrogenic, isotonic, clear solution of atropine sulfate in water for injection with sodium chloride sufficient to render the solution isotonic. Each mL contains atropine sulfate, 0.4 mg; benzyl alcohol, 9 mg; sodium chloride 9 mg; and may contain sulfuric acid for pH adjustment, pH 3.5 (3.0 to 3.8).
  Atropine sulfate injection will be supplied in multidose vials containing 20 mL.
  Each vial will only be used to administer a single dose, to a single subject.
  Interventions: Drug: Atropine Sulphate Injection

INTERVENTIONS:
Drug: Atropine Sulfate Ophthalmic Solution — Atropine sulfate ophthalmic solution, USP 1% is a sterile topical anti-muscarinic indicated for cyclopegia, mydriasis, and penalization of the healthy eye in the treatment of amblyopia. Each mL of Atropine Sulfate Ophthalmic Solution USP, 1% contains active ingredient: atropine sulfate 10 mg equivalent to 8.3 mg of atropine. Inactive ingredients include benzalkonium chloride 0.1 mg (0.01%), dibasic sodium phosphate, edetate disodium, hypromellose (2910), monobasic sodium phosphate, hydrochloric acid and/or sodium hydroxide may be added to adjust pH (3.5 to 6.0), and water for injection, USP.
  Arms: High Dose Sublingual; Low Dose Sublingual
Drug: Atropine Sulphate Injection — Atropine sulfate injection, USP, 8mg/20mL (0.4 mg per mL) is a sterile, nonpyrogenic, isotonic, clear solution of atropine sulfate in water for injection with sodium chloride sufficient to render the solution isotonic. Each mL contains atropine sulfate, 0.4 mg; benzyl alcohol, 9 mg; sodium chloride 9 mg; and may contain sulfuric acid for pH adjustment, pH 3.5 (3.0 to 3.8).
  Arms: Intravenous (IV)

SUMMARY:
This randomized, three-sequence, three-period, phase 1 study is designed to assess the bioavailability and pharmacokinetics (PK) of sublingually administered atropine sulfate ophthalmic solution 1% USP (at 0.5 mg and 1.0 mg; test) compared to atropine sulfate injection administered IV (1.0 mg; reference).

DETAILED DESCRIPTION:
This is a randomized, three-sequence, three-period crossover study to assess the bioavailability and PK of a single dose of atropine administered sublingually in healthy adult volunteers. At least 15 healthy male and female volunteers will be enrolled to obtain approximately 12 evaluable subjects in the per protocol population. Eligible subjects will be randomized at a 1:1:1 ratio to receive one of three treatment dosing sequences (A, B, or C).

Subjects assigned to treatment dosing sequence A will receive a low dose sublingually at Visit 1; Day 1 (Period 1), a high dose sublingually at Visit 2; Day 8 (Period 2) and an IV dose at Visit 3; Day 15 (Period 3).

Subjects assigned to treatment dosing sequence B will receive a high dose sublingually at Visit 1; Day 1 (Period 1), an IV dose at Visit 2; Day 8 (Period 2) and a low dose sublingually at Visit 3; Day 15 (Period 3).

Subjects assigned to treatment dosing sequence C will receive an IV dose at Visit 1; Day 1 (Period 1), a low dose sublingually at Visit 2; Day 8 (Period 2), and a high dose sublingually at Visit 3; Day 15 (Period 3).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and nonpregnant female volunteers between the ages of 18 and 55 years at time of randomization
2. Willing and able to provide written informed consent
3. Females who are of childbearing potential and are sexually active with a male partner must have used an acceptable method of birth control for at least 2 months prior to Screening, and must agree to continue using an acceptable method of birth control from Screening to Follow-up (Day 21).

   A female of childbearing potential is defined as postonset menarche and premenopausal female capable of becoming pregnant. This does not include females who meet any of the following conditions: menopausal > 2 years, tubal ligation > 1 year, bilateral salpingo-oophorectomy, or hysterectomy.

   Adequate contraception is defined as a contraceptive method with a failure rate of less than 1% per year when used consistently and correctly and when applicable, in accordance with the product label. Examples include oral contraceptives, injectable progestogen, implants of etonogestrel or levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, intrauterine device or intrauterine system, or male partner sterilization at least 6 months prior to the female subject's Screening Visit.
4. In the judgment of the investigator, the subject is in good health, based on review of medical history and the results of screening evaluation (including vital signs, physical examination, 12-lead ECG, and routine clinical laboratory testing, performed no more than 14 days prior to randomization into the study)
5. Able to comply with the dosing instructions and available to complete the study Schedule of Events

Exclusion Criteria:

1. Females who have a positive pregnancy test or who are breastfeeding
2. Subjects with thyroid disease as evidenced by a thyroid-stimulating hormone (TSH) < 0.9 × lower limit of normal (LLN) or > 1.2 × upper limit of normal (ULN) at screening. (This test will not be repeated prior to subsequent dosing.)
3. Subjects with aspartate aminotransferase (AST), alanine aminotransferase (ALT), or serum creatinine > 1.5 × ULN at screening. (These tests will not be repeated prior to subsequent dosing.)
4. Have known human immunodeficiency virus (HIV), or acute or chronic hepatitis B or hepatitis C infection based on medical history; or test positive for any of these at Screening. Subjects who have been effectively treated for hepatitis C, as evidenced by a negative hepatitis C ribonucleic acid (RNA) confirmation test and who no longer require antiviral therapy, are eligible for participation. (Screening tests will not be repeated prior to subsequent dosing.)
5. Subjects who took any prescription medications (with the exception of oral contraceptives or hormone replacement therapy) within 30 days of screening. Prior to each dose, the investigator will review prohibited medication use and determine whether the subject should be terminated from further dosing.
6. Subjects who took any over-the-counter medication/vitamins/herbal supplements in the last 72 hours prior to screening. Prior to each dose, the investigator will review prohibited medication use and determine whether the subject should be terminated from further dosing.
7. Subjects with glaucoma and/or history of ocular surgery (including Lasik), ocular trauma, or congenital ocular disorder
8. Subjects with any history of heart disease including but not limited to coronary artery disease, arrhythmia (treated or untreated), congestive heart failure, pacemaker, history of vasovagal syncope, peripheral vascular disease, or claudication
9. Subjects with clinically significant arrhythmias or abnormal conduction; abnormal conduction is defined as a prolonged PR or QRS, or a QTc ≥ 450 msec for males or ≥ 470 msec for females
10. Subjects with a history of partial organic pyloric stenosis, chronic constipation, or other gastrointestinal motility issue
11. Subjects with a history of xerostomia due to an underlying disease or previous radiation therapy to the head and neck
12. Males with history of symptomatic prostatic hypertrophy; males or females with a history of hesitancy or retention
13. Subjects with a blood pressure > 140/90 mm Hg taken after the subject has been seated and resting for at least five minutes
14. Subjects with a history or current diagnosis of myasthenia gravis
15. Subjects with a history of drug or alcohol abuse in the last two years or evidence of a positive urine drug test at screening. (This screening test will not be repeated prior to subsequent dosing.)
16. Subjects with a known sensitivity or prior adverse reaction to atropine

Subjects cannot be rescreened for exclusionary laboratory test results. Potentially exclusionary vital sign results may be repeated once. If a subject's repeat vitals remain exclusionary or the investigator determines that the repeat vital signs could pose a risk to the subject participating in the study, then the subject will be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-04 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schwartz, MD MPH, Study Chair — Department of Health and Human Services
Locations (1):
- High Point Clinical Trials Center, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajpal S, Ali R, Bhatnagar A, Bhandari SK, Mittal G. Clinical and bioavailability studies of sublingually administered atropine sulfate. Am J Emerg Med. 2010 Feb;28(2):143-50. doi: 10.1016/j.ajem.2008.10.025. PMID 20159382
- [Background] Pai S, Ghezzi EM, Ship JA. Development of a Visual Analogue Scale questionnaire for subjective assessment of salivary dysfunction. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Mar;91(3):311-6. doi: 10.1067/moe.2001.111551. PMID 11250628

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence A: Low Dose Sublingual - High Dose Sublingual - IV: Subjects assigned to treatment dosing sequence A will receive a low dose sublingually at Visit 1; Day 1 (Period 1), a high dose sublingually at Visit 2; Day 8 (Period 2) and an IV dose at Visit 3; Day 15 (Period 3).
- Sequence B: High Dose Sublingual - IV - Low Dose Sublingual: Subjects assigned to treatment dosing sequence B will receive a high dose sublingually at Visit 1; Day 1 (Period 1), an IV dose at Visit 2; Day 8 (Period 2) and a low dose sublingually at Visit 3; Day 15 (Period 3).
- Sequence C: IV - Low Dose Sublingual - High Dose Sublingual: Subjects assigned to treatment dosing sequence C will receive an IV dose at Visit 1; Day 1 (Period 1), a low dose sublingually at Visit 2; Day 8 (Period 2), and a high dose sublingually at Visit 3; Day 15 (Period 3).
Period: Period 1 (Visit 1; Day 1)
Arm/Group | Sequence A: Low Dose Sublingual - High Dose Sublingual - IV | Sequence B: High Dose Sublingual - IV - Low Dose Sublingual | Sequence C: IV - Low Dose Sublingual - High Dose Sublingual
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0
Period: Period 2 (Visit 2; Day 8)
Arm/Group | Sequence A: Low Dose Sublingual - High Dose Sublingual - IV | Sequence B: High Dose Sublingual - IV - Low Dose Sublingual | Sequence C: IV - Low Dose Sublingual - High Dose Sublingual
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0
Period: Period 3 (Visit 3; Day 15)
Arm/Group | Sequence A: Low Dose Sublingual - High Dose Sublingual - IV | Sequence B: High Dose Sublingual - IV - Low Dose Sublingual | Sequence C: IV - Low Dose Sublingual - High Dose Sublingual
Started | 5 | 4 | 5
Completed | 5 | 4 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population includes all participants who were randomized and received at least 1 study drug dose.
Groups:
- A: Low Dose Sublingual - High Dose Sublingual - IV: Subjects assigned to treatment dosing sequence A will receive a low dose sublingually at Visit 1; Day 1 (Period 1), a high dose sublingually at Visit 2; Day 8 (Period 2) and an IV dose at Visit 3; Day 15 (Period 3).
- B: High Dose Sublingual - IV - Low Dose Sublingual: Subjects assigned to treatment dosing sequence B will receive a high dose sublingually at Visit 1; Day 1 (Period 1), an IV dose at Visit 2; Day 8 (Period 2) and a low dose sublingually at Visit 3; Day 15 (Period 3).
- C: Intravenous (IV)-Low Dose Sublingual-High Dose Sublingual: Subjects assigned to treatment dosing sequence C will receive an IV dose at Visit 1; Day 1 (Period 1), a low dose sublingually at Visit 2; Day 8 (Period 2), and a high dose sublingually at Visit 3; Day 15 (Period 3).
- Total: Total of all reporting groups
Arm/Group | A: Low Dose Sublingual - High Dose Sublingual - IV | B: High Dose Sublingual - IV - Low Dose Sublingual | C: Intravenous (IV)-Low Dose Sublingual-High Dose Sublingual | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 5 | 15
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (7.46) | 29.2 (5.76) | 35.0 (3.87) | 33.8 (6.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 3 | 7
  Male | 5 | 1 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 4 | 5 | 4 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 3 | 8
  White | 1 | 2 | 2 | 5
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 5 | 15
Body Mass Index [Median (Full Range); unit: kg/m^2] — Body mass index, calculated as: Weight (kg) / Height (m)2
  kg/m^2 | 24.76 [21.1 to 29.7] | 25.16 [21.2 to 35.2] | 34.13 [26.8 to 39.0] | 29.55 [21.1 to 39.0]
Screening Xerostomia Assessment - Difficulty Swallowing (0-10) [Mean (Standard Deviation); unit: Scores on a scale] — Subject reported xerostomia score of difficulty swallowing due to mouth dryness, assessed by questionnaire previously validated for measurement of salivary gland dysfunction. Xerostomia scores were based on a scale of 0 to 10, with 0 being not difficult at all and 10 being very difficult.
  Scores on a scale | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Screening Xerostomia Assessment - Dryness of Lips (0-10) [Mean (Standard Deviation); unit: Scores on a scale] — Subject reported xerostomia score of dryness of lips, assessed by questionnaire previously validated for measurement of salivary gland dysfunction. Xerostomia scores were based on a scale of 0 to 10, with 0 being not dry at all and 10 being very dry.
  Scores on a scale | 0.4 (0.55) | 1.6 (2.07) | 0.2 (0.45) | 0.7 (1.33)
Screening Xerostomia Assessment - Dryness of Tongue (0-10) [Mean (Standard Deviation); unit: Scores on a scale] — Subject reported xerostomia score of dryness of tongue, assessed by questionnaire previously validated for measurement of salivary gland dysfunction. Xerostomia scores were based on a scale of 0 to 10, with 0 being not dry at all and 10 being very dry.
  Scores on a scale | 0 (0) | 0 (0) | 0 (0) | 0 (0)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve to From Time Zero to Infinity (AUC_∞)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 2, 4, 6, 10, 15, 20, 30, 45, and 60 minutes, and 2, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using the noncompartmental method for extravascular (for sublingual doses) or IV infusion routes of administration.
  AUC_∞ is summarized by study dosage as the geometric mean and coefficient of variation of the geometric mean for all evaluable participants and expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model.
Time Frame: Pre-dose through 8 hours post-dose at Days 1, 8 and 15
Population: The PK analysis population includes all subjects who were randomized, received at least 1 study drug dose, and have PK samples collected for the applicable period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Groups:
- Low Dose Sublingual; High Dose Sublingual: Atropine sulfate ophthalmic solution, USP 1% is a sterile topical anti-muscarinic indicated for cyclopegia, mydriasis, and penalization of the healthy eye in the treatment of amblyopia. Each mL of Atropine Sulfate Ophthalmic Solution USP, 1% contains active ingredient: atropine sulfate 10 mg equivalent to 8.3 mg of atropine.
- Intravenous: Atropine sulfate injection is indicated for temporary blockade of severe or life-threatening muscarinic effects, e.g., as an antisialagogue, an antivagal agent, an antidote for organophosphorus, carbamate, or muscarinic mushroom poisoning, and to treat symptomatic bradycardia.
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 11 | 14 | 14
min*ng/mL | 286.396 (26.6) | 493.808 (27.3) | 816.465 (22.0)
Statistical Analysis 1: Comparison: Low Dose Sublingual vs High Dose Sublingual; Test type: Other — Estimation only; Mixed Models Analysis; Geometric ratio of least-square means = 0.579, 90% CI 2-sided [0.5265 to 0.6360] — Only subjects who had at least 2 periods where study drug was received with an evaluable PK profile were included in the comparisons
Statistical Analysis 2: Comparison: Low Dose Sublingual vs Intravenous; Test type: Other — Estimation only; Mixed Models Analysis; Geometric ratio of least-square means = 0.349, 90% CI 2-sided [0.3171 to 0.3839] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: High Dose Sublingual vs Intravenous; Test type: Other — Estimation only; Mixed Models Analysis; Geometric ratio of least-square means = 0.603, 90% CI 2-sided [0.5524 to 0.6582] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Timepoint (AUC_t)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 2, 4, 6, 10, 15, 20, 30, 45, and 60 minutes, and 2, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using the noncompartmental method for extravascular (for sublingual doses) or IV infusion routes of administration.
  AUC_t is summarized by study dosage as the geometric mean and coefficient of variation of the geometric mean for all evaluable participants and expressed as min*ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model.
Time Frame: Pre-dose through 8 hours post-dose at Days 1, 8 and 15
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: min*ng/mL
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 14 | 15 | 14
min*ng/mL | 218.195 (20.2) | 408.061 (23.9) | 717.665 (23.2)
Statistical Analysis 1: Comparison: Low Dose Sublingual vs High Dose Sublingual; Test type: Other — Estimation only; Mixed Models Analysis; Geometric ratio of least-square means = 0.546, 90% CI 2-sided [0.4971 to 0.6004] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Low Dose Sublingual vs Intravenous; Test type: Other — Estimation only; Mixed Models Analysis; Geometric ratio of least-square means = 0.306, 90% CI 2-sided [0.2788 to 0.3367] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: High Dose Sublingual vs Intravenous; Test type: Other — Estimation only; Mixed Models Analysis; Geometric ratio of least-square means = 0.561, 90% CI 2-sided [0.5104 to 0.6164] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Concentration (C_max)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 2, 4, 6, 10, 15, 20, 30, 45, and 60 minutes, and 2, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using the noncompartmental method for extravascular (for sublingual doses) or IV infusion routes of administration.
  C_max is summarized by study dosage as the geometric mean and coefficient of variation of the geometric mean for all evaluable participants and expressed as ng/mL. Geometric ratios of least-square means and associated 90% confidence intervals are reported from a linear mixed model.
Time Frame: Pre-dose through 8 hours post-dose at Days 1, 8 and 15
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 14 | 15 | 14
ng/mL | 0.883 (27.2) | 1.639 (30.5) | 18.247 (66.9)
Statistical Analysis 1: Comparison: Low Dose Sublingual vs High Dose Sublingual; Test type: Other — Estimation only; Mixed Models Analysis; Geometric ratio of least-square means = 0.549, 90% CI 2-sided [0.4273 to 0.7118] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Low Dose Sublingual vs Intravenous; Test type: Other — Estimation only; Mixed Models Analysis; Geometric ratio of least-square means = 0.049, 90% CI 2-sided [0.0381 to 0.0641] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: High Dose Sublingual vs Intravenous; Test type: Other — Estimation only; Mixed Models Analysis; Geometric ratio of least-square means = 0.090, 90% CI 2-sided [0.0695 to 0.1167] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Time to Maximum Concentration (t_max)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 2, 4, 6, 10, 15, 20, 30, 45, and 60 minutes, and 2, 4, 6, and 8 hours. PK parameters were estimated for each subject and sublingual dosing period using the noncompartmental method. This outcome is not applicable for the intravenous dosing period.
  t_max is summarized by study dosage as the mean and standard deviation for all evaluable participants and expressed as minutes.
Time Frame: Pre-dose through 8 hours post-dose at Days 1, 8 and 15
Population: The PK analysis population includes all subjects who were randomized, received at least 1 study drug dose, and have PK samples collected for the applicable periods for extravascular (sublingual) routes of administration. Note: t_max was not applicable to intravenous dosing.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 14 | 15 | 0
Minutes | 125.4 (69.81) | 107.1 (47.78) |

5. Primary Outcome: Terminal Elimination Half-Life (t_1/2)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 2, 4, 6, 10, 15, 20, 30, 45, and 60 minutes, and 2, 4, 6, and 8 hours. PK parameters were estimated for each subject and period using the noncompartmental method for extravascular (for sublingual doses) or IV infusion routes of administration.
  t_1/2 is summarized by study dosage as the mean and standard deviation for all evaluable participants and expressed as minutes.
Time Frame: Pre-dose through 8 hours post-dose at Days 1, 8 and 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Intravenous (IV): Atropine sulfate injection is indicated for temporary blockade of severe or life-threatening muscarinic effects, e.g., as an antisialagogue, an antivagal agent, an antidote for organophosphorus, carbamate, or muscarinic mushroom poisoning, and to treat symptomatic bradycardia.
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous (IV)
Number analyzed (Participants) | 11 | 14 | 14
Minutes | 176.187 (75.0887) | 171.258 (49.9828) | 179.327 (60.412)

6. Primary Outcome: Volume of Distribution (V_d/F)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 2, 4, 6, 10, 15, 20, 30, 45, and 60 minutes, and 2, 4, 6, and 8 hours. PK parameters were estimated for each subject and sublingual dosing period using the noncompartmental method. This outcome is not applicable for the intravenous dosing period.
  V_d/F is summarized by study dosage as the mean and standard deviation for all evaluable participants and expressed as liters.
Time Frame: Pre-dose through 8 hours post-dose at Days 1, 8 and 15
Population: The PK analysis population includes all subjects who were randomized, received at least 1 study drug dose, and have PK samples collected for the applicable periods for extravascular (sublingual) routes of administration. Note: V_d/F is not applicable to intravenous dosing.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 11 | 14 | 0
L | 423.71 (119.774) | 496.70 (138.811) |

7. Primary Outcome: Clearance (CL/F)
Description: Blood samples to measure atropine plasma concentrations were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 2, 4, 6, 10, 15, 20, 30, 45, and 60 minutes, and 2, 4, 6, and 8 hours. PK parameters were estimated for each subject and sublingual dosing period using the noncompartmental method. This outcome is not applicable for the intravenous dosing period.
  CL/F is summarized by study dosage as the mean and standard deviation for all evaluable participants and expressed as mL/min.
Time Frame: Pre-dose through 8 hours post-dose at Days 1, 8 and 15
Population: The PK analysis population includes all subjects who were randomized, received at least 1 study drug dose, and have PK samples collected for the applicable periods for extravascular (sublingual) routes of administration. Note: CL/F is not applicable to intravenous dosing.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 11 | 14 | 0
mL/min | 1800.800 (473.3604) | 2098.806 (632.8211) |

8. Secondary Outcome: Treatment-Emergent Adverse Events
Description: Number of patients with treatment-emergent adverse events
Time Frame: Day 1 through Day 21
Population: The Safety population includes all subjects who were randomized and received at least 1 study drug dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 14 | 15 | 14
Participants | 1 | 1 | 4

9. Secondary Outcome: Treatment-Emergent Serious Adverse Events
Description: Number of patients with treatment-emergent serious adverse events
Time Frame: Day 1 through Day 21
Population: The Safety population includes all subjects who were randomized and received at least 1 study drug dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 14 | 15 | 14
Participants | 0 | 0 | 0

10. Secondary Outcome: Xerostomia Assessment - Difficulty Swallowing Due to Mouth Dryness
Description: Subject reported xerostomia scores were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 10, 20, 30, 40, 50, and 60 minutes. Scores were assessed by questionnaire (0-10 point scale, with 0 being not difficult at all and 10 being very difficult) previously validated for measurement of salivary gland dysfunction.
  The maximum xerostomia score representing difficulty swallowing due to mouth dryness was calculated for each subject and dose. Maximum xerostomia scores were summarized by study dosage as the mean and standard deviation.
Time Frame: Pre-dose through 1 hour post-dose at Days 1, 8 and 15
Population: The Safety population includes all subjects who were randomized and received at least 1 study drug dose.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 14 | 15 | 14
Scores on a scale | 0.3 (1.07) | 0.3 (0.82) | 2.0 (2.77)

11. Secondary Outcome: Xerostomia Assessment - Dryness of Lips
Description: Subject reported xerostomia scores were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 10, 20, 30, 40, 50, and 60 minutes. Scores were assessed by questionnaire (0-10 point scale, with 0 being not dry at all and 10 being very dry) previously validated for measurement of salivary gland dysfunction.
  The maximum xerostomia score representing dryness of lips was calculated for each subject and dose. Maximum xerostomia scores were summarized by study dosage as the mean and standard deviation.
Time Frame: Pre-dose through 1 hour post-dose at Days 1, 8 and 15
Population: The Safety population includes all subjects who were randomized and received at least 1 study drug dose.
Measure: Mean (Standard Deviation); unit: Maximum Score
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 14 | 15 | 14
Maximum Score | 1.1 (1.38) | 1.5 (1.85) | 2.9 (2.88)

12. Secondary Outcome: Xerostomia Assessment - Dryness of Tongue
Description: Subject reported xerostomia scores were collected during each dosing visit at the following time points: time 0 (predose), and postdose at 10, 20, 30, 40, 50, and 60 minutes. Scores were assessed by questionnaire (0-10 point scale, with 0 being not dry at all and 10 being very dry) previously validated for measurement of salivary gland dysfunction.
  The maximum xerostomia score representing dryness of tongue was calculated for each subject and dose. Maximum xerostomia scores were summarized by study dosage as the mean and standard deviation.
Time Frame: Pre-dose through 1 hour post-dose at Days 1, 8 and 15
Measure: Mean (Standard Deviation); unit: Maximum Score
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
Number analyzed (Participants) | 14 | 15 | 14
Maximum Score | 0.3 (0.61) | 0.3 (0.46) | 2.1 (2.67)

ADVERSE EVENTS:
Time Frame: AEs were collected from the time of consent until completion of the follow-up period after the last administration of study drug Follow-up (Day 21).
Description: Events grade 1 or higher were be recorded on the appropriate AE electronic case report form (eCRF) for this study.
  The study site graded the severity of AEs experienced by the study participants according to the criteria set forth in the NCI-CTCAE Version 5.0.
Arm/Group | Low Dose Sublingual | High Dose Sublingual | Intravenous
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 1/15 | 4/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Sublingual (N=14) | High Dose Sublingual (N=15) | Intravenous (N=14)
Abdominal Pain - Lower (Gastrointestinal disorders) | 1 (1) | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 (1) | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2 (2)
Dizziness (Nervous system disorders) | 0 | 0 | 1 (1)
Headache (Nervous system disorders) | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/39/NCT04290039/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/39/NCT04290039/ICF_001.pdf